CLINICAL TRIAL: NCT05234645
Title: Short Term Effects of Probiotics in the Human Micro-vascular Physiology - Comparison Between Older and Younger Healthy, Sedentary Adults: a Pilot Study.
Brief Title: Short Term Effects of Probiotics in the Human Micro-vascular Physiology
Acronym: PIMCO-KEFIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ER5560941
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Microcirculation; Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Younger group (Experimental): Fifteen participants, between 18 and 35 years of age. Participants are not pregnant; are healthy and suffering from no chronic diseases with the potential to influence vascular function; non-smoker; sedentary (defined via the completion of the international physical activity questionnaire; IPAQ); and were not consuming regularly probiotic-containing products. Additionally, a medical questionnaire was completed to exclude anyone with overt chronic disease.
  Interventions: Other: Kefir consumption
- Older group (Experimental): Fourteen participants, between 55 and 75 years of age. Participants are not pregnant; are healthy and suffering from no chronic diseases with the potential to influence vascular function; non-smoker; sedentary (defined via the completion of the international physical activity questionnaire; IPAQ); and were not consuming regularly probiotic-containing products. Additionally, a medical questionnaire was completed to exclude anyone with overt chronic disease.
  Interventions: Other: Kefir consumption

INTERVENTIONS:
Other: Kefir consumption — Following confirmation of eligibility and the provision of informed consent, recruited participants were provided with a 4-week supply of kefir (Live Kefir Company, Pontefract, UK) being instructed to consume 150ml of Kefir per day for the whole 4-week period. No break periods of kefir consumption were offered to any of the participants. In addition, they were instructed to not change their usual dietary habits and exercise routine for the study duration.

SUMMARY:
While the beneficial properties of kefir consumption have been thoroughly studied for many years, very little research has been conducted to explore the potential protective properties of kefir consumption to the endothelium in humans. Therefore, the aim of the current study is to explore the short-term efficacy of kefir consumption in improving endothelial function in older and younger healthy, sedentary adults.

ELIGIBILITY:
Inclusion Criteria:

All recruited participants were either 18-35 yrs. or 55-75 yrs.

Exclusion Criteria:

Pregnancy; chronic diseases with the potential to influence vascular function; smoking status; sedentary (defined via the completion of the international physical activity questionnaire; IPAQ); regular consumption of probiotic-containing products; any overt chronic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Microcirculatory function | Baseline.
  Skin blood flow will be measured as cutaneous red blood cell flux using a Laser Doppler Flowmeter (LDF). Local thermal hyperaemia will be induced using a heating disc surrounding the probe. The probe will be attached to the skin using a double-sided adhesion sticker. Participants will be rested in a supine position in a temperature-controlled room with a constant ambient temperature of 24° C for 35 minutes. Baseline skin blood flow data will be recorded for 5 minutes with the local heating disc temperature set at 30° C. Following this, rapid local heating will be initiated to obtain maximal vasodilation and the temperature will be increased by 1° C every 10 seconds until 42° C was reached. This will then be maintained for 30 minutes following, which the test will be completed.
Microcirculatory function | 8 weeks.
  Skin blood flow will be measured as cutaneous red blood cell flux using a Laser Doppler Flowmeter (LDF). Local thermal hyperaemia will be induced using a heating disc surrounding the probe. The probe will be attached to the skin using a double-sided adhesion sticker. Participants will be rested in a supine position in a temperature-controlled room with a constant ambient temperature of 24° C for 35 minutes. Baseline skin blood flow data will be recorded for 5 minutes with the local heating disc temperature set at 30° C. Following this, rapid local heating will be initiated to obtain maximal vasodilation and the temperature will be increased by 1° C every 10 seconds until 42° C was reached. This will then be maintained for 30 minutes following, which the test will be completed.

SECONDARY OUTCOMES:
Anthropometry - 1 | Baseline.
  Stature, waist and hip circumferences will be measured (all in cms).
Anthropometry - 1 | 8 weeks.
  Stature, waist and hip circumferences will be measured (all in cms).
Anthropometry - 2 | Baseline.
  Body mass will be measured.
Anthropometry - 2 | 8 weeks.
  Body mass will be measured.
SF-IPAQ | Baseline.
  The SF-IPAQ questionnaire will be completed, to assess physical activity levels.
A discontinuous, sub-maximal test, coupled with transcutaneous oxygen pressure (TcPO2). | Baseline
  A discontinuous, sub-maximal test, involving four rounds of exercise will measure the participants' transcutaneous oxygen pressure (TcPO2).TcPO2 values will be measured and recorded by a sensor. Measurements will be taken, using a TINA TCM400 TcPO2 device (Radiometer, Copenhagen, Denmark). The electrode will be placed on the participants' back, below the right scapula. The testing protocol includes a total of 20 min on a cycle ergometer (Monark894E, Vansbro, Sweden) with a 2-min break after each 5 min of exercise. Participants will maintain a speed of 80 revolutions per minute, and after each 5-min period, an extra 0.2 kg of resistance will be added to the ergometer, with a 1 kg of starting resistance value. Participants will be encouraged to reach their maximum exertion limit before completing the assessment but could stop before the end of the test if they feel so.
A discontinuous, sub-maximal test, coupled with transcutaneous oxygen pressure (TcPO2). | 8 weeks.
  A discontinuous, sub-maximal test, involving four rounds of exercise will measure the participants' transcutaneous oxygen pressure (TcPO2).TcPO2 values will be measured and recorded by a sensor. Measurements will be taken, using a TINA TCM400 TcPO2 device (Radiometer, Copenhagen, Denmark). The electrode will be placed on the participants' back, below the right scapula. The testing protocol includes a total of 20 min on a cycle ergometer (Monark894E, Vansbro, Sweden) with a 2-min break after each 5 min of exercise. Participants will maintain a speed of 80 revolutions per minute, and after each 5-min period, an extra 0.2 kg of resistance will be added to the ergometer, with a 1 kg of starting resistance value. Participants will be encouraged to reach their maximum exertion limit before completing the assessment but could stop before the end of the test if they feel so.
Blood pressure | Baseline.
  Diastolic and systolic blood pressure will be recorded from the left arm at 5-minute intervals throughout the protocol (Dinamap Dash 2500, GE Healthcare, USA).
Blood pressure | 8 weeks.
  Diastolic and systolic blood pressure will be recorded from the left arm at 5-minute intervals throughout the protocol (Dinamap Dash 2500, GE Healthcare, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Markos Klonizakis, D.Phil, Principal Investigator — Reader (Clinical Physiology)
Locations (1):
- Sheffield Hallam University, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No